CLINICAL TRIAL: NCT05396417
Title: Early Recovery After Surgery for Patients Undergoing Cesarean Delivery; Adherence to the Institutional Guideline
Brief Title: How Well do the Current Cesarean Deliveries Adhere to the Published ERAS Guidelines?
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Women's Hospital HUS (Other)
Responsible Party: Principal Investigator, Antti Vaananen, Principal investigator, Women's Hospital HUS
Other Study IDs: Tutkimussuunnitelma25032022_I
Record Dates: First submitted 2022-05-27; First posted 2022-05-31 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cesarean delivery: Any urgency any reason
  Interventions: Procedure: cesarean delivery

INTERVENTIONS:
Procedure: cesarean delivery — Cesarean delivery under any form of anesthesia for any reason and for any indication

SUMMARY:
Local guidelines for the postoperative care of women who have undergone cesarean delivery at the HUS/Women's hospital are based recommendations by the ERAS society. This study will take a prospective sample of 500 parturients who have gone through a cesarean delivery and their care will be verified against the local check-list for cesarean delivery.

DETAILED DESCRIPTION:
The study will produce a snapshot of the current state of treatment in the third largest delivery hospital in Europe. The study will include cesarean deliveries in all urgency categories.

The data will be collected prospectively by enrolling parturients in consecutive order from the study start date. The data will be collected in the form of a paper check list that is to be filled up by the nursing staff and doctors who are taking care of the parturient through her stay at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for ERAS protocol cesarean delivery
* Cesarean delivery for any indication
* Any anesthesia method
* Any urgency category

Exclusion Criteria:

* Age under 18 years

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Women undergoing cesarean delivery at the University of Helsinki central hospital/Women's hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Level of adherence to the ERAS guidelines after elective or emergency cesarean delivery | 3 days post surgery
  To which extent does the postoperative treatment of the parturients meet the ERAS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- HUS/Women's hospital dept of obstetrics, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No